CLINICAL TRIAL: NCT00653029
Title: An fMRI Study of Selective Attention, Working Memory, and Effort After Mild Traumatic Brain Injury
Brief Title: An fMRI Study of Attention and Effort After Concussion
Status: Terminated | Type: Observational
Why Stopped: Difficulties with recruitment and MRI scanner became unavailable.
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Brian Rieger, Chief Psychologist PM&R, State University of New York - Upstate Medical University
Other Study IDs: 5406
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Post Concussive Syndrome
Keywords: Post concussion syndrome; Mild traumatic brain injury; Effort; fmri
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens
Oversight: Data Monitoring Committee: No

SUMMARY:
Approximately 1.1 million people a year suffer a mild traumatic brain injury (MTBI), or concussion, in the United States. Although most MTBI patients fully recover, as many as 28% have physical, cognitive, and/or emotional symptoms up to 6 months post-injury. When symptoms persist past three months, it is known as post-concussion syndrome (PCS). The cause of PCS is unknown, as structural neuroimaging and neuropsychological (NP) testing results are often normal. However, recent functional magnetic resonance imaging (fMRI) research in concussed adults showed differences in brain activity compared to controls on working memory tasks, despite normal structural MRI and neuropsychological findings. We propose improving this research by assessing brain activation patterns during simple versus complex attention and working memory tasks in 10 concussed adults via fMRI. This will be the first study to examine brain activation patterns associated with the degree of effort applied to testing, a factor known to confound interpretation of NP test performance. Validated computerized measures of selective attention (Modified Stroop Interference Task), working memory (n-back), and effort (Green's Medical Symptom Validity Test; MSVT) will be used. Ten paid controls will be used for comparative purposes. We hypothesize that concussed patients will show less brain activation than controls on complex versus simple working memory tasks and that activation patterns in concussed patients will generally be lower in those with suboptimal effort. We will also characterize self-reported emotional and physical symptoms in the PCS patients, which has not been done in prior fMRI research with this population.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI (based on criteria of the American Congress of Rehabilitation Medicine)
* Aged 18 to 60
* History of non-penetrating head injury
* Obtaining medical assistance (e.g., personal physician, Emergency Room) within 24 hours post-injury

Exclusion Criteria:

* No prior history of prior post-concussion syndrome (i.e, uncomplicated mild TBI)
* Moderate to severe TBI
* Substance dependence
* Learning disorder
* Attention-deficit disorder
* Mental retardation
* Severe psychiatric disorder requiring hospitalization
* Previous central nervous system disease
* Absence of neurosurgery
* No evidence of alcohol/drug use related to the injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
BOLD Response | Patients will undergo fMRI at least one month after injury
  Blood Oxygen Level Dependent Response protocol on fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Dominic A Carone, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States